CLINICAL TRIAL: NCT04549051
Title: Percutaneous Interruption of the Coracohumeral Ligament for the Treatment of Frozen Shoulder.
Acronym: CHLTenex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2020-11998
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Adhesive Capsulitis
MeSH Terms: conditions — Bursitis | interventions — Anesthetics, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Tenex plus local anesthetic (Experimental): Use of the TENEX device for sectioning of the CHL
  Interventions: Device: Tenex; Drug: Local anesthetic
- Local Anesthetic (Other): Only Local anesthetic will be injected into the CHL. This arm will have the option to cross over into Tenex arm at 1 month
  Interventions: Drug: Local anesthetic

INTERVENTIONS:
Device: Tenex — Local anesthetic plus Tenex into the coracohumeral ligament for adhesive capsulitis
  Arms: Tenex plus local anesthetic
Drug: Local anesthetic — Only local anesthetic into the coracohumeral ligament for adhesive capsulitis

SUMMARY:
Percutaneous Interruption of the Coracohumeral Ligament for the treatment of Frozen Shoulder.

DETAILED DESCRIPTION:
Chronic inflammation of the shoulder joint capsule and its associated structures can lead to clinically significant symptoms, including insidious onset of pain, and ultimately restricting range of motion. Although the underlying mechanism for adhesive capsulitis (AC) is not well defined, some studies suggest that fibroblast proliferation and thickening of the coracohumeral ligament (CHL) is a proposed mechanism for which AC and subsequent prolonged immobilization and symptoms present (1, 2, 3). Other studies suggest that it is due to a combination of capsular fibrosis and inflammation within the synovium, and other focus on the fact that thickening of the CHL is responsible for limiting external rotation in patients affected by adhesive capsulitis (1).

AC coined frozen shoulder by Codman in 1934 [2), has an estimated prevalence of 2-3% in the general population, with ages 40-70 affected most commonly, and predominantly women. While the precise etiology remains undefined, it can be secondary to trauma or an idiopathic etiology and has been found to have an incidence as high as 20% in diabetic patients, with worse functional outcomes when compared to non-diabetic patients. Hypothyroidism and cerebrovascular disease have also been shown to be associated with an increased risk of developing AC (4). AC is typically a clinical diagnosis. However, both magnetic resonance and ultrasonography have consistently shown thickening of the CHL (1). Several studies have compared arthrographic evidence of findings in adhesive capsulitis, and many reported a thickening of the CHL in cases of frozen shoulder as compared to control subjects (2). In a study implementing shear-wave elastography (SWE), the CHL in patients diagnosed with adhesive capsulitis was thicker and stiffer (4).

Interventions aimed at improving AC and CHL damage, clinical symptomatology, as well as histopathological findings range from rest and physical therapy, local injections and hydrodilation, to advanced surgical interventions (4, 5). These surgical options include manipulation under anesthesia (MUA) and arthroscopic capsulotomy. MUA is an aggressive mobilization of the joint in an effort to lyse adhesions and to stretch the contracted glenohumeral capsule. Despite potential benefits, MUA has been associated with superior labral anterior and posterior (SLAP) lesions, bankart lesions, capsular tears, hemarthrosis, and even humeral or glenoid fractures (4). Arthroscopic capsulotomy allows for direct visualization of the CHL and confirmation of the diagnosis of AC, and several studies have shown improvement in pain relief as well as range of motion (4). However, patients who did not benefit from this intervention were women, typically over the age of 50, with a past medical history of diabetes mellitus. CHL resection has also been described as a potential treatment option for AC (6, 7), with current therapy limited to a surgical approach. Management of refractory disease through arthroscopic capsular release has been shown to improve pain and increase range-of-motion (8, 9, 4). A sequela of arthroscopic surgery is postoperative persistent AC, which some surgeons attempt to prophylactically prevent with adequate postoperative pain control so that the patient can participate in a physical therapy program. The potential limitations of current conservative management and IRB NUMBER: 2020-11998 IRB APPROVAL DATE: 11/17/2020 sequelae of surgical approaches have prompted additional novel therapies. International have researchers developed an ultrasound guided technique with a scalpel incision of the CHL to address this need. Scalpel use is not the standard of care for interventional musculoskeletal pain treatments and our team decided to improve this limitation. Blades and scalpels limit US visibility, thus marginalizing the safety of the procedure. Our team used a percutaneous, ultrasound visible, needle shaped, tissue cutting device to lesion the CHL while improving upon the potential safety concerns. The tool, TENEX®, is widely used by Pain physicians to perform percutaneous tenotomies and has been described in the management of various tendinous pathologies (10, 11, 12, 13, 14, 15).; this device was selected because the gross architectural similarities of tendon and ligament suggest that the CHL could be modified by this tool. Our novel procedure was performed on cadavers to provide proof of concept

The authors performed cadaveric dissection in 8 cadaveric shoulders with the hypothesis that sonographically guided percutaneous dissection will result in sectioning of the coracohumeral ligament. In this study we found that complete sectioning was reproducibly achieved in 7 minutes with approximately 250 passes of the device. This was the desired outcome for improving the shoulder ROM (16). This shows proof of concept and we want to perform this procedure in living subjects for validation. If the results are positive patients can have an outpatient procedure in the interventional pain clinic with desirable results. This cadaveric technique study has already been submitted to Pain Medicine journal for publication.

In addition to the above proof of concept above this procedure was performed in living subjects. A peer reviewed paper was submitted based on data from these subjects. 7 patients were selected for the publication as these patients had follow-ups as requested by the reviewer. In these patients the average improvement in external rotation was 40 degrees and the average abduction improvement was 31 degrees. All patients retained this improvement in shoulder ROM at follow-up visits. Of note, one patients follow-up visit was 116 after the procedure and her improvement in ROM was 60 and 110 in external rotation and abduction respectively. Given these outcomes the authors decided to do a prospective RCT.

ELIGIBILITY:
Inclusion Criteria:

* Established Diagnosis of Adhesive capsulitis (AC) Ligament Flavum >3mm, diagnosed by US evaluation decreased shoulder ROM in external rotation and abduction (50% of unaffected side)
* Patients who have tried other conventional therapies like steroid treatments, surgical treatments, physiotherapy with little (defined by less than 20 degrees improvement in shoulder ROM - external rotation) to no improvement in the shoulder ROM

Exclusion Criteria:

* Age less than 18 years and greater than 89 years
* Patients with AC but showing improvement in shoulder ROM progressively (defined by improvement in ROM > 200 external rotation or 20 degrees per week when undergoing physiotherapy)
* Patients who are currently pregnant

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2023-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sayed Wahezi, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu CH, Chen WS, Wang TG. Elasticity of the Coracohumeral Ligament in Patients with Adhesive Capsulitis of the Shoulder. Radiology. 2016 Feb;278(2):458-64. doi: 10.1148/radiol.2015150888. Epub 2015 Aug 31. PMID 26323030
- [Background] Mengiardi B, Pfirrmann CW, Gerber C, Hodler J, Zanetti M. Frozen shoulder: MR arthrographic findings. Radiology. 2004 Nov;233(2):486-92. doi: 10.1148/radiol.2332031219. Epub 2004 Sep 9. PMID 15358849
- [Background] Dias R, Cutts S, Massoud S. Frozen shoulder. BMJ. 2005 Dec 17;331(7530):1453-6. doi: 10.1136/bmj.331.7530.1453. PMID 16356983
- [Background] Le HV, Lee SJ, Nazarian A, Rodriguez EK. Adhesive capsulitis of the shoulder: review of pathophysiology and current clinical treatments. Shoulder Elbow. 2017 Apr;9(2):75-84. doi: 10.1177/1758573216676786. Epub 2016 Nov 7. PMID 28405218
- [Background] Maund E, Craig D, Suekarran S, Neilson A, Wright K, Brealey S, Dennis L, Goodchild L, Hanchard N, Rangan A, Richardson G, Robertson J, McDaid C. Management of frozen shoulder: a systematic review and cost-effectiveness analysis. Health Technol Assess. 2012;16(11):1-264. doi: 10.3310/hta16110. PMID 22405512
- [Background] Hagiwara Y, Sekiguchi T, Ando A, Kanazawa K, Koide M, Hamada J, Yabe Y, Yoshida S, Itoi E. Effects of Arthroscopic Coracohumeral Ligament Release on Range of Motion for Patients with Frozen Shoulder. Open Orthop J. 2018 Sep 18;12:373-379. doi: 10.2174/1874325001812010373. eCollection 2018. PMID 30288192
- [Background] Yukata K, Goto T, Sakai T, Fujii H, Hamawaki J, Yasui N. Ultrasound-guided coracohumeral ligament release. Orthop Traumatol Surg Res. 2018 Oct;104(6):823-827. doi: 10.1016/j.otsr.2018.01.016. Epub 2018 Mar 19. PMID 29567320
- [Background] Austgulen OK, Oyen J, Hegna J, Solheim E. [Arthroscopic capsular release in treatment of primary frozen shoulder]. Tidsskr Nor Laegeforen. 2007 May 17;127(10):1356-8. Norwegian. PMID 17519989
- [Background] Chen SK, Chien SH, Fu YC, Huang PJ, Chou PH. Idiopathic frozen shoulder treated by arthroscopic brisement. Kaohsiung J Med Sci. 2002 Jun;18(6):289-94. PMID 12355929
- [Background] Sanchez PJ, Grady JF, Saxena A. Percutaneous Ultrasonic Tenotomy for Achilles Tendinopathy Is a Surgical Procedure With Similar Complications. J Foot Ankle Surg. 2017 Sep-Oct;56(5):982-984. doi: 10.1053/j.jfas.2017.06.015. PMID 28842108
- [Background] Kamineni S, Butterfield T, Sinai A. Percutaneous ultrasonic debridement of tendinopathy-a pilot Achilles rabbit model. J Orthop Surg Res. 2015 May 20;10:70. doi: 10.1186/s13018-015-0207-7. PMID 25986341
- [Background] Chimenti RL, Stover DW, Fick BS, Hall MM. Percutaneous Ultrasonic Tenotomy Reduces Insertional Achilles Tendinopathy Pain With High Patient Satisfaction and a Low Complication Rate. J Ultrasound Med. 2019 Jun;38(6):1629-1635. doi: 10.1002/jum.14835. Epub 2018 Oct 2. PMID 30280399
- [Background] Barnes DE, Beckley JM, Smith J. Percutaneous ultrasonic tenotomy for chronic elbow tendinosis: a prospective study. J Shoulder Elbow Surg. 2015 Jan;24(1):67-73. doi: 10.1016/j.jse.2014.07.017. Epub 2014 Oct 8. PMID 25306494
- [Background] Koh JS, Mohan PC, Howe TS, Lee BP, Chia SL, Yang Z, Morrey BF. Fasciotomy and surgical tenotomy for recalcitrant lateral elbow tendinopathy: early clinical experience with a novel device for minimally invasive percutaneous microresection. Am J Sports Med. 2013 Mar;41(3):636-44. doi: 10.1177/0363546512470625. Epub 2013 Jan 9. PMID 23302261
- [Background] Zhu J, Hu B, Xing C, Li J. Ultrasound-guided, minimally invasive, percutaneous needle puncture treatment for tennis elbow. Adv Ther. 2008 Oct;25(10):1031-6. doi: 10.1007/s12325-008-0099-6. PMID 18791678
- [Background] Homsi C, Bordalo-Rodrigues M, da Silva JJ, Stump XM. Ultrasound in adhesive capsulitis of the shoulder: is assessment of the coracohumeral ligament a valuable diagnostic tool? Skeletal Radiol. 2006 Sep;35(9):673-8. doi: 10.1007/s00256-006-0136-y. Epub 2006 May 25. PMID 16724200

RESULTS

PARTICIPANT FLOW:
Groups:
- Local Anesthetic First Then Tenex Plus Local Anesthetic: Local anesthetic injected into the CHL. Patients in this arm also had the option to cross over into Tenex plus Local Anesthetic arm at 1 month (~4 weeks).
  Procedure Description:
  Local anesthetic: Local anesthetic into the coracohumeral ligament for adhesive capsulitis
  Tenex: Local anesthetic plus Tenex into the coracohumeral ligament for adhesive capsulitis
- Tenex Plus Local Anesthetic Alone: Use of the TENEX device for sectioning of the CHL
  Procedure Description:
  Tenex: Local anesthetic plus Tenex into the coracohumeral ligament for adhesive capsulitis
  Local anesthetic: Local anesthetic into the coracohumeral ligament for adhesive capsulitis
Period: First Intervention (4 Weeks)
Arm/Group | Local Anesthetic First Then Tenex Plus Local Anesthetic | Tenex Plus Local Anesthetic Alone
Started | 16 | 30
Completed | 16 (Follow-up Duration was one month for local anesthetic group. All 16 Subjects completed their one month follow-up period without any adverse events. 9 out of 16 subjects crossed over into TENEX group after their one-month follow-up. Remaining 7 subjects monitored only for adverse events.) | 30 (Follow-up Duration was one year for TENEX group. All 30 Subjects completed their one month follow-up period and continued to be monitored for one year.)
Not Completed | 0 | 0
Period: Optional Second Intervention (11 Months)
Arm/Group | Local Anesthetic First Then Tenex Plus Local Anesthetic | Tenex Plus Local Anesthetic Alone
Started | 9 (9 of 16 subjects crossed over into TENEX group after their one-month follow-up. Remaining 7 subjects only monitored for adverse events. Of these 7 subject, 5 had Adverse Events (4 SAEs and 1 AE) and 2 were lost to follow up) | 30
Completed | 9 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Local Anesthetic First Then Tenex Plus Local Anesthetic: Only Local anesthetic injected into the CHL. Patients in this arm had the option to cross over into Tenex plus Local Anesthetic arm at 1 month (~4 weeks).
  Procedure Description:
  Local anesthetic: Local anesthetic into the coracohumeral ligament for adhesive capsulitis
  Tenex: Local anesthetic plus Tenex into the coracohumeral ligament for adhesive capsulitis
- Total: Total of all reporting groups
Arm/Group | Tenex Plus Local Anesthetic Alone | Local Anesthetic First Then Tenex Plus Local Anesthetic | Total
Number analyzed (Participants) | 26 | 13 | 39
Age, Customized [Mean (Standard Deviation); unit: years] | 65.00 (11.59) | 56.00 (11.93) | 62.21 (11.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 11 | 31
  Male | 6 | 2 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 26 | 13 | 39
BMI [Mean (Standard Deviation); unit: kg/m^2] | 36.34 (6.88) | 30.45 (5.78) | 32.18 (6.47)
Affected Arm (Right/Left) [Number; unit: participants] — The affected arm (Ieft or right) of each patient is noted.
  participants
    Left Arm | 13 | 4 | 17
    Right Arm | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Range of Motion of the Shoulder
Description: Change in shoulder range of motion (ROM) (external rotation and abduction) procedure by at least 100%, measured with goniometer. Increased degrees of motion is indicative of more favorable/better outcomes.
Time Frame: Immediately following procedure, up to 60 minutes
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Tenex Plus Local Anesthetic Alone | Local Anesthetic First Then Tenex Plus Local Anesthetic
Number analyzed (Participants) | 26 | 13
degrees
  External Rotation | 61 (18) | 49 (16)
  Abduction | 80 (14) | 64 (13)

2. Secondary Outcome: Durability of Local Anesthetic - Change in Range Of Motion (ROM)
Description: Shoulder abduction and external rotation measured with goniometer. Increased degrees of motion is indicative of more favorable/better outcomes.
Time Frame: Baseline (Before the procedure) and at 1 month
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Local Anesthetic First Then Tenex Plus Local Anesthetic
Number analyzed (Participants) | 13
degrees
  External Rotation at Baseline (Before the procedure) | 29 (8)
  External Rotation at 1-Month | 32 (7)
  Abduction at Baseline (Before the procedure) | 53 (15)
  Abduction at 1-Month | 57 (14)

3. Secondary Outcome: Durability of the TENEX - Change in Range Of Motion (ROM)
Description: as for outcome 2
Time Frame: Immediately after the procedure and at the long term follow-up (10 months to 2 years)
Population: In addition to 26 subjects in the TENEX group, 9 Subjects in Control group were crossed over into the TENEX arm at their 1-month visit.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Tenex Plus Local Anesthetic Alone
Number analyzed (Participants) | 35
degrees
  External Rotation Immediately after the procedure | 63 (17)
  External Rotation in the long term | 62 (18)
  Abduction Immediately after the procedure | 78 (15)
  Abduction in the long term | 77 (21)

4. Secondary Outcome: Change of Pain Intensity Score for Local Anesthetic Group
Description: Measured by visual analog scale (VAS). VAS is a validated, subjective measure for for acute and chronic pain. Range of possible values: 0-10. (Higher score indicates more pain)
Time Frame: at the Baseline visit (Before the procedure) and at the 1-month visit
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Local Anesthetic First Then Tenex Plus Local Anesthetic
Number analyzed (Participants) | 13
score on a scale
  VAS at baseline | 8 [7 to 8]
  VAS at 1-month | 8 [7.75 to 8.25]

5. Secondary Outcome: Change of Pain Intensity Score for TENEX Group
Description: as for outcome 4
Time Frame: at the Baseline visit (before the procedure) and at the long-term follow-up (10 months to 2 years)
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Tenex Plus Local Anesthetic Alone
Number analyzed (Participants) | 35
score on a scale
  VAS at baseline | 8 [8 to 9]
  VAS at long term (10 months to 2 years) | 3 [2 to 7]

6. Secondary Outcome: Change of the Oxford Shoulder Score for Local Anesthetic Group
Description: Measured by The Oxford Shoulder Score (OSS) questionnaire form. The Oxford Shoulder Score (OSS) is a 12-item patient-report questionnaire with a 0-4 scoring format, developed to identify functional changes of the shoulder. Range of possible values: 0-48. (Higher score represents a better outcome)
Time Frame: at the baseline (before the procedure) and at the 1-month visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Local Anesthetic First Then Tenex Plus Local Anesthetic
Number analyzed (Participants) | 13
score on a scale
  at the baseline | 10.8 (7.9)
  at the 1-month | 13.8 (8.2)

7. Secondary Outcome: Change of the Oxford Shoulder Score for TENEX Group
Description: as for outcome 6
Time Frame: at the baseline (before the procedure) and at the long term follow-up (10 months to 2 years)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tenex Plus Local Anesthetic Alone
Number analyzed (Participants) | 35
score on a scale
  at the baseline | 7.4 (4.6)
  at the long term (10 months to 2 years) | 31.8 (11.7)

ADVERSE EVENTS:
Time Frame: Each patient was followed for adverse events from the date of enrollment into the study until the date of their last follow-up, approximately 1 year.
Groups:
- Tenex Plus Local Anesthetic Alone: Use of the TENEX device for sectioning of the CHL
  There were 30 subjects directly enrolled to TENEX group and 1 out of these 30 subjects had SAE.
  After 9 Subjects' crossing over, there were totally 39 subject who got the TENEX procedure in this group.
  3 out of 9 crossed over subjects had SAE after crossing over. So, totally 4 subjects had SAE after receiving the TENEX procedure.
  Procedure Description:
  Tenex: Local anesthetic plus Tenex into the coracohumeral ligament for adhesive capsulitis Local anesthetic: Only local anesthetic into the coracohumeral ligament for adhesive capsulitis
- Local Anesthetic First Then Tenex Plus Local Anesthetic: Only Local anesthetic injected into the CHL. This arm had the option to cross over into Tenex arm at 1 month.
  There were 16 subjects enrolled to Local Anesthetic group. 9 Subjects crossed over into TENEX group at the one month follow-up.
  So after 1 month follow-up, Only 7 Subjects remained in Local Anesthetic group and these 7 subjects did not have any SAE.
  3 out of 9 crossed over subjects had SAE after crossing over.
  Procedure Description:
  Local anesthetic: Only local anesthetic into the coracohumeral ligament for adhesive capsulitis
Arm/Group | Tenex Plus Local Anesthetic Alone | Local Anesthetic First Then Tenex Plus Local Anesthetic
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/16
Serious Adverse Events (participants affected / at risk) | 4/30 | 0/16
Other Adverse Events (participants affected / at risk) | 1/30 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenex Plus Local Anesthetic Alone (N=30) | Local Anesthetic First Then Tenex Plus Local Anesthetic (N=16)
Serious Adverse Event (Surgical and medical procedures) | 4 (4) | 0 (0) — Subject underwent the reverse shoulder arthroplasty on the effected (study) site
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenex Plus Local Anesthetic Alone (N=30) | Local Anesthetic First Then Tenex Plus Local Anesthetic (N=16)
Shoulder Trauma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Shoulder trauma which was not related to study procedures

LIMITATIONS AND CAVEATS:
This study represents a small population of patients with a CHL-related ROM deficit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT04549051/Prot_SAP_ICF_000.pdf